CLINICAL TRIAL: NCT01455935
Title: Wake up Symptomatic Stroke in Acute Brain Ischemia (WASSABI) Trial
Brief Title: Wake up Symptomatic Stroke - Benefit of Intravenous Clot Busters or Endovascular Intervention
Acronym: WASSABI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jacobs Neurological Institute (Other)
Collaborators: University at Buffalo Neurosurgery (Other); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Tareq Kass-Hout, Chief Vascular/Neurology Resident in charge of stroke, Jacobs Neurological Institute
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: NEU 3200411A
Record Dates: First submitted 2011-10-07; First posted 2011-10-20 (Estimated); Last update posted 2012-03-30 (Estimated); Status verified 2012-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Tissue Plasminogen Activator

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Medical Therapy (Active Comparator): Current standard of care per the latest stroke guidelines
  * Permissive Hypertension up to 220
  * Antipletelets therapy:
    1. ASA 81 mg PO daily or
    2. Plavix 75 mg PO daily or
    3. Aggrenox 225mg PO twice daily
  * Anti-inflammatory therapy:
    1. Lipitor 80 mg PO daily or
    2. Crestor 20 mg PO daily
  Interventions: Drug: Anti-platelets and statin
- Intravenous Thrombolysis (Experimental): Full dose Intravenous thrombolysis
  * 0.9 mg/kg
  * Maximum dose is 90 mg
  * 10% of the dose will be given over one minute
  * 90% of the dose will be infused over 1 hour
  * Admission to Neuro Intensive Care Unit(NICU) for 24 hours if no complications
  * Neuro checks every 5 minutes during the infusion
  * Neuro checks every hour after the infusion for 24 hours
  Interventions: Drug: alteplase
- Intra-Arterial Therapy (Experimental): -Choice of therapy per experienced Endovascular surgeon and includes:
  1. Intra arterial Activase (Maximum dose of 22 mg)
  2. MERCI device (Maximum of 3 tries per device, no standard time frame for how long the procedure takes)
  3. PENUMBRA device (no standard time frame for how long the procedure takes)
  Interventions: Procedure: intra arterial intervention

INTERVENTIONS:
Drug: Anti-platelets and statin
  Arms: Medical Therapy
Drug: alteplase — Full dose Intravenous thrombolysis
  * 0.9 mg/kg
  * Maximum dose is 90 mg
  * 10% of the dose will be given over one minute
  * 90% of the dose will be infused over 1 hour
  * Admission to Neuro Intensive Care Unit(NICU) for 24 hours if no complications
  * Neuro checks every 5 minutes during the infusion
  * Neuro checks every hour after the infusion for 24 hours
  Arms: Intravenous Thrombolysis
Procedure: intra arterial intervention — 1. Intra arterial Activase (Maximum dose of 22 mg)
  2. MERCI device (Maximum of 3 tries per device, no standard time frame for how long the procedure takes)
  3. PENUMBRA device (no standard time frame for how long the procedure takes)
  Arms: Intra-Arterial Therapy

SUMMARY:
The purpose of the trial is to study the safety and the effectiveness of using CT Perfusion studies as an indicator to treat stroke patients with unknown time of onset.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria: To be eligible for entry into this study, candidates must meet all of the following eligibility criteria at the time of Emergency Department presentation:

1. Age: 18-80 years old
2. Ischemic Wake Up Stroke (Unknown time of onset but less than 24 hours since last seen normal)
3. National Institute of Health Stroke Scale (NIHSS) 8-22
4. Evidence of penumbra on Computed Tomography Perfusion(CTP) as mentioned above
5. Alberta Stroke Program Early Computed Tomography (CT) Score (ASPECTS 7 or more)
6. Signed informed consent

Exclusion Criteria:

Exclusion Criteria: Potential study patients will be excluded from study entry if any of the following exclusion criteria exist at the time of screening:

1. Evidence of intracranial hemorrhage (Intracerebral hematoma, intraventricular hemorrhage, subarachnoid hemorrhage (SAH), epidural hemorrhage, acute or chronic subdural hematoma (SDH)) on the baseline CT
2. Historical Modified Rankin Scale (mRS) of ≥2
3. National Institute of Health Stroke Scale (NIHSS)<8 at the time of treatment
4. Positive pregnancy test in women at age of childbearing
5. Intracranial or intraspinal surgery within 3 months
6. Stroke or serious head injury within 3 months
7. History of intracranial hemorrhage
8. Uncontrolled hypertension at time of treatment (eg, >185 mm Hg systolic or >110 mm Hg diastolic)
9. Seizure at the onset of stroke
10. Active internal bleeding
11. Intracranial neoplasm
12. Arteriovenous malformation or aneurysm
13. Clinical presentation suggesting post-MI pericarditis
14. Known bleeding diathesis including but not limited to current use of oral anticoagulants producing an Internation normalized ratio (INR) >1.7
15. Internation normalized ratio (INR) >1.7
16. Administration of heparin within 48 hours preceding the onset of stroke with an elevated activated Partial Thromboplastin Time(aPTT) at presentation
17. Platelet count <100,000/mm
18. Major surgery within 2 weeks
19. GastroIntestinal (GI) or urinary tract hemorrhage within 3 weeks
20. Aggressive treatment required to lower blood pressure
21. Glucose level <50 or >400 mg/dL
22. Arterial puncture at a noncompressible site or lumbar puncture within 1 week

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-12 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale (mRS) | 90 days
  Modified Rankin Scale (mRS) 90 days post treatment

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) | 24 hour
  National Institute of Health Stroke Scale (NIHSS) 24 hours post treatment.
National Institute of Health Stroke Scale (NIHSS) | 3-29 day
  National Institute of Health Stroke Scale (NIHSS) at discharge (3-29 days)
Modified Rankin Scale (mRS) | 30 post treatment
  Modified Rankin Scale (mRS) at 30 days post treatment
Thrombolysis In Myocardial Infarction (TIMI) Flow | Pre - up to1 hour prior to procedure and post will be up to1 hour after completion of procedure
  Thrombolysis In Myocardial Infarction (TIMI) flow pre and post the intervention as an indicator of revascularization rate
Thomboylsis in Cerebral Ischemia (TICI) flow | Pre - will be no more than 1 hour prior to procedure and post will be no more then 1 hour after completion of procedure
  Thomboylsis in Cerebral Ischemia (TICI) flow pre and post intervention as an indicator of revascularization rate
symptomatic intracranial Hemorrhage (ICH) | 72 hours
  Incidence of symptomatic symptomatic intracranial Hemorrhage (ICH) within 72 hours of intervention defined by ECASSIII as 4 points worsening in NIHSS
National Institute of Health Stroke Scale (NIHSS) | 30 Days
  at 30 Day visit National Institute of Health Stroke Scale (NIHSS) will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Elad I Levy, MD, Study Director — University at Buffalo Neurosurgery; Tareq Kass-Hout, MD, Principal Investigator — Jacobs Neurological Institute
Locations (1):
- Millard Fillmore Gates Circle Hospital, Buffalo, New York, United States